CLINICAL TRIAL: NCT00131469
Title: A Study to Assess the Effectiveness of Teriparatide (FORTEO) for Increasing Bone Mass and Improving Bone Strength in Adults Affected With Osteogenesis Imperfecta (OI)
Brief Title: Study of Teriparatide (FORTEO) to Treat Adults With Osteogenesis Imperfecta
Acronym: OI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Eli Lilly and Company (Industry); Osteogenesis Imperfecta Foundation (Other); National Institutes of Health (NIH) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Eric Orwoll, MD, Professor Of Medicine, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IBMD-OI; UL1RR024140 (NIH)
Record Dates: First submitted 2005-08-16; First posted 2005-08-18 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Osteogenesis Imperfecta
Keywords: Osteogenesis Imperfecta; Brittle Bone Disease; Fragility Fractures
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teriparatide (FORTEO) (Active Comparator): Once daily SQ administration of Teriparatide (FORTEO) 20 ug for 18 months
  Interventions: Drug: Teriparatide (FORTEO)
- Placebo (Placebo Comparator): Daily SQ placebo for 18 months
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Teriparatide (FORTEO) — Teriparatide (FORTEO) 20mcg, subcutaneous injection, once daily
  Other Names: FORTEO
  Arms: Teriparatide (FORTEO)
Drug: Placebos
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness of teriparatide (FORTEO), which is human parathyroid hormone 1-34, for increasing bone mass and improving bone structure in adults affected with Osteogenesis Imperfecta (OI).

DETAILED DESCRIPTION:
The purpose of this study is to determine the effectiveness of teriparatide (FORTEO), which is human parathyroid hormone 1-34, for increasing bone mass and improving bone structure in adults affected with Osteogenesis Imperfecta (OI). Osteogenesis imperfecta is an inherited disorder of type I collagen, a major component of bones, and is characterized by multiple fractures and deformities. OI affects approximately 1-2 of every 10,000 individuals. Virtually all of the studies of potential treatments for OI have evaluated the effects of medications only on children with OI. There is no cure for osteogenesis imperfecta and there is no established medical therapy for adults with the disorder. There are very limited data concerning the usefulness of parathyroid hormone therapy in OI. An effective anabolic therapy for the treatment of adult patients with OI could be a valuable asset to the affected patients. In this study, the working hypothesis is that individuals affected with OI who are treated with Forteo will experience increased spine and hip bone mineral density and an increase in bone strength. Although Forteo is not expected to change the defect in the collagen produced, but is postulated to increase the quantity of bone formed and improve bone strength.

This will be a placebo controlled, double blinded trial; half the patients will receive Forteo 20 ug/day SQ. Adult patients (age at least 18 yrs) with OI will be enrolled for a treatment duration of 18 months. Blood, urine, and bone density/strength tests will be done during the study to assess efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Previous established diagnosis of Osteogenesis Imperfecta AND
* > 2 previous adult fractures, AND/OR
* BMD at lumbar spine, femoral neck or total hip T score < -2.0

Exclusion Criteria:

* Open epiphyses.
* History of external beam radiation to the skeleton.
* Pagets disease.
* Bone metastases or skeletal malignancies.
* Total lifetime exposure to any antiresorptive medication < 90 days (Primary Inclusion).
* Treatment with any antiresorptive medication 12 months proceeding enrollment - (Secondary Inclusion).
* Women with OI who are pregnant or unwilling to use 1 form of contraception.
* Vitamin D insufficiency (25-hydroxyvitamin D <15ng/ml)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2005-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric S Orwoll, M.D., Principal Investigator — Oregon Health and Science University; Jay Shapiro, M.D., Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.; Brendan Lee, M.D., PhD, Principal Investigator — Balor College of Medicine; Sandra Veith, CRA, Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (3):
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Oregon Health & Science University, Portland, Oregon
  - Baylor College of Medicine, Department of Molecular and Human Gentics, Houston, Texas

REFERENCES:
- [Derived] Orwoll ES, Shapiro J, Veith S, Wang Y, Lapidus J, Vanek C, Reeder JL, Keaveny TM, Lee DC, Mullins MA, Nagamani SC, Lee B. Evaluation of teriparatide treatment in adults with osteogenesis imperfecta. J Clin Invest. 2014 Feb;124(2):491-8. doi: 10.1172/JCI71101. Epub 2014 Jan 27. PMID 24463451
- See also: Osteogenesis Imperfecta Foundation — http://oif.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was formally enrolled but then dropped out before the first study treatment was administered.
Groups:
- Placebo: Daily SQ placebo for 18 months
  Placebos
Period: Overall Study
Arm/Group | Teriparatide (FORTEO) | Placebo
Started | 38 | 40
Completed | 29 | 27
Not Completed | 9 | 13
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Protocol Violation | 3 | 1
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — scan not analyzable | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide (FORTEO) | Placebo | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (12.9) | 41.2 (10.1) | 41 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 16 | 16 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Spine Bone Mineral Density (BMD)
Description: bone density by dual energy xray absorptiometry
Time Frame: baseline and 18 months
Measure: Mean (Standard Error); unit: percentage of change in g/cm2
Arm/Group | Teriparatide (FORTEO) | Placebo
Number analyzed (Participants) | 29 | 27
percentage of change in g/cm2 | 6.1 (1.5) | 2.8 (1.3)

2. Secondary Outcome: Total Hip BMD
Description: bone density by dual energy xray absorptiometry
Time Frame: baseline and 18 months
Measure: Mean (Standard Error); unit: percentage of change in g/cm2
Arm/Group | Teriparatide (FORTEO) | Placebo
Number analyzed (Participants) | 22 | 26
percentage of change in g/cm2 | 2.6 (2) | -2.4 (1.8)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Teriparatide (FORTEO) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 1/40
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 0/38 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No